CLINICAL TRIAL: NCT04837118
Title: PancStrength: Safety, Feasibility, and Acceptability of a Tele-Exercise Resistance Training Intervention During Pancreatic Cancer Treatment
Brief Title: Resistance Training Intervention to Improve Physical Function in Patients With Pancreatic Cancer Receiving Combination Chemotherapy or Have Undergone Surgery, PancStrength Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0147; NCI-2021-02028 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0147 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (resistance training) (Experimental): SEE DETAILED DESCRIPTION.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Educational Intervention — Receive handouts containing dietary recommendations
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Participate in a resistance training program
  Other Names: Strength Training

SUMMARY:
This clinical trial studies the safety of a real-time tele-exercise resistance training (training done using a tablet) in maintaining skeletal muscle, strength, physical function, and health-related quality of life in patients with pancreatic cancer who are receiving combination chemotherapy or have undergone surgery for the treatment of pancreatic cancer. Tele-exercise resistance training may improve physical function and quality of life in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety of a progressive, home-based, tele-exercise resistance training (tele-RT) intervention in patients undergoing first line FOLFIRINOX chemotherapy for advanced pancreatic ductal adenocarcinoma (PDAC) (Study 1) and in survivors who have undergone pancreatic cancer resection (Study 2).

SECONDARY OBJECTIVES:

I. Evaluate the feasibility and acceptability of the tele-RT intervention.

II. Evaluate changes in the following exploratory outcome measures over the course of first-line FOLFIRINOX for advanced PDAC and associations between resistance training (RT) volumes and their changes:

IIa. Muscular strength IIb. Muscular endurance IIc. Body composition (skeletal muscle mass) IId. Aerobic fitness IIe. Self-reported physical activity IIf. Self-reported physical functioning IIg. Fatigue IIh. Peripheral neuropathy IIi. Health-related quality of life (QOL) IIj. Completion of intended chemotherapy dose (Among patients who are undergoing chemotherapy; all participants in Study 1 and some in Study 2) IIk. Exercise motivation IIl. Exercise self-efficacy IIm. Social support for exercise IIn. Reduction or change in FOLFIRINOX treatment plan III. Evaluate cancer care providers' (treating physicians and other clinical personnel) perspectives regarding the feasibility and acceptability of the tele-RT intervention for their patients.

OUTLINE:

STUDY 1: During the first 2-3 months of first line FOLFIRINOX chemotherapy, patients complete at least 4 tele-RT sessions over 30-45 minutes each, every 2 weeks. Patients receive handouts created by MD Anderson Cancer Center (MDACC) clinical dietitians including individualized recommendations for daily protein intake and information about healthy protein supplementation during chemotherapy. Patient may also attend a visit with a registered dietician (or delegate dietician) per standard of care, if they have renal insufficiency, special dietary needs, or difficulty adhering to protein recommendations.

STUDY 2: After standard of care surgical resection, patients complete at least 4 tele-RT sessions over 30-45 minutes each, every 2 weeks for 2-3 months. Patients receive handouts created by MDACC clinical dietitians including individualized recommendations for daily protein intake and information about healthy protein supplementation during chemotherapy. Patient may also attend a visit with a registered dietician (or delegate dietician) per standard of care, if they have renal insufficiency, special dietary needs, or difficulty adhering to protein recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven pancreatic adenocarcinoma, advanced stage (III-IV) (study 1) OR biopsy-proven pancreatic adenocarcinoma, at least 10 weeks post-surgical tumor resection and currently with no radiographic evidence of disease on recent computerized tomography (CT) scan (study 2)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Treatment plan of first-line FOLFIRINOX chemotherapy with planned return visit to MD Anderson Main Campus for restaging (study 1) OR plans to return to MDACC for restaging appointments in 3-4 months, including follow up CT scan (study 2)
* Able to schedule baseline (T0) appointment for fitness testing and program teaching at the Behavioral Research and Treatment Center (BRTC) or able to schedule remote fitness testing and program teaching
* Able to understand the description of the study, exercise program, and willing to participate
* Home access to wireless internet (Wi-Fi) and agreement to engage with study personnel for real-time tele-RT sessions
* Age >= 18
* Meet all screening requirements
* PROVIDERS (FOR ACCEPTABILITY INTERVENTION): All GI medical oncologists, GI surgeons, advanced practice providers, and clinical dietitians who are involved in participants' care and have some interaction with intervention personnel during recruitment, referral, scheduling, or follow up will be asked to complete questionnaires assessing intervention acceptability. The exact number of providers who will be asked to complete questionnaires will depend on whether patients enroll from the different GI Medical Oncology and GI Surgery clinics, but we expect 10-20 providers to be eligible

Exclusion Criteria:

* Non-English speaking
* Has participated in regular RT (RT for all major muscle groups at least twice per week) throughout the month prior to recruitment
* Unable to complete the baseline assessment questionnaires or functional assessments
* Screen failure for exercise safety based on Physical Activity Readiness Questionnaire (PAR-Q) and/or Patient Reported Outcomes Measurement Information System (PROMIS) questions
* Underlying unstable cardiac or pulmonary disease or symptomatic cardiac disease (New York Heart Association functional class III or IV)
* Recent fracture or acute musculoskeletal injury that precludes the ability to weight bear fully on all 4 limbs in order to participate in an exercise intervention
* Numeric pain rating scale of >= 7 out of 10
* Myopathic or rheumatologic disease that impacts physical function
* FEMALES ONLY: Known pregnancy, as communicated to study personnel by clinicians in gastrointestinal (GI) Medical Oncology; females of childbearing potential receive advice to use methods of contraception per usual care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the tele-resistance training (RT) program | 3-4 months
  Safety will be assessed based on the rate of musculoskeletal injuries and other adverse health events that participants incur while participating in tele-RT sessions. Participants will be monitored throughout the exercise intervention for musculoskeletal injuries and other adverse health events and referred to a Physical Medicine and Rehabilitation physician or their gastrointestinal (GI) Medical Oncology teams as necessary. The association of the injury with strength training will be assessed by asking participants to rate the injury on a scale of 1-4 (1=not related, 2=unlikely related, 3=likely related, 4=definitely related). The severity of the injury will be rated on a scale of 1-4 (1=mild/no change in daily activity, 2=some limitation of daily activity, 3=major limitation of daily activity, 4=life threatening). The duration for which daily activities were impacted will be rated on a scale from 1-5 (1=no change, 2=1-3 days, 3=4-7 days, 4=1-2 weeks, 5=more than 2 weeks).
Post-exercise muscle soreness | 3-4 months
  Soreness will be assessed at the beginning of each tele-RT session, with participants asked to describe how soreness has changed since the previous RT session and how soreness has changed over the course of RT sessions. If soreness is not becoming more manageable with ongoing RT, participants will be referred to Dr. Ngo-Huang (study co-principal investigator [PI] and physiatrist) for follow-up to rule out any underlying injuries.
Body composition | 3-4 months
  Cross-sectional areas (CSA) of skeletal muscle, intramuscular fat, visceral fat, and subcutaneous fat will be measured using SliceOMatic software (TomoVision, 2012) using computed tomography images routinely obtained for cancer assessment and staging purposes. Imaging dates will align with cancer staging and restaging appointments at T0 and T1. Cross-sectional areas at the L3 vertebral level will be standardized to the square of participants' heights in meters. Average radiodensity (in Hounsfield Units) of skeletal muscle will also be collected using SliceOMatic software.
Aerobic fitness | 3-4 months
  Will be measured using 6-minute walk test (6MWT) distance, measured in meters. For participants who undergo remote exercise testing, the 2-minute step test will be used to assess aerobic fitness. Participants will be guided to step in place as quickly as possible, raising each knee to the proper height (midway between the opposite knee and hip), with trainers recording the number of complete steps they can complete in 2 minutes.

SECONDARY OUTCOMES:
Acceptability for Feasibility | 3-4 months
  Will be assessed with the following variables: 1)Uptake rate: Study enrollment will be considered feasible if 70% of eligible patients who are approached to consider study enrollment actually consent and enroll. 2) Study completion rate: If 70% of participants who complete T0 measures (fitness and survey measures) also complete measures at T1. 3) Tele-RT session attendance rate: If the rate of session completion is >= 70%. 4) Adherence to prescribed exercise volume (sets x repetitions x resistance): If the volume of exercise completed is >= 70% of the volume prescribed.
Acceptability for participants | 3-4 months
  Assessed with the Participant Evaluation of Feasibility and Acceptability questionnaire, adapted from Ingram, et al (2010). This questionnaire includes both Likert Scale and open-ended questions. Likert Scale items will be rated on 5-point scales (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree). Acceptability will be assessed on an item-by-item basis and as an average item score, with scores >= 4 ("agree" to "strongly agree") indicating acceptability. Responses to open-ended questions will be analyzed qualitatively to inform development of further iterations of the exercise intervention. Qualitative analysis will follow a content analysis strategy to systematically define units of text, quantify them, and group them into meaningful categories.
Acceptability for providers | 3-4 months
  Assessed with a brief program evaluation questionnaire distributed to all GI medical oncologists, GI surgeons, advanced practice providers, and clinical dietitians who are involved in participants' care and have some interaction with intervention personnel during recruitment, referral, scheduling, or follow up. Provider acceptability questionnaires will be distributed via REDCap immediately following collection of T1 data from the final study participant and will include Likert Scale items and open-ended items adapted from the Participant Evaluation of Feasibility and Acceptability.
Dynamic upper- and lower-body muscular strength | 3-4 months
  Strength in upper- and lower-body muscle groups will be measured using the following 1-repetition maximum (1RM) lifts: chest press, seated row, leg press, and leg extension. 1RM tests are considered the gold standard for assessing muscular strength in non-laboratory situations. 1RM tests are defined as the maximal weight that can be lifted once with correct lifting technique and are used by athletic trainers, health and fitness professionals and rehabilitation specialists to assess strength and to evaluate training programs. They will be performed in the following sequence, ordered from largest to smallest muscle groups and alternating between upper and lower body movements to allow for sufficient rest: leg press, chest press, leg extension, seated row.
Dynamic upper- and lower-body muscular endurance | 3-4 months
  Endurance of upper and lower body muscle groups as measured by the maximum number of repetitions performed at 70% of the T0 1RM for each of the following lifts: leg press, chest press, leg extension, seated row. Participants will rest sufficiently between movements and will perform tests in the same order that they performed 1RM testing. Participants who undergo remote enrollment and exercise testing will undergo the following exercise "field tests" to assess muscular strength and endurance: 1) 30-second chair stand test (to assess lower body strength and muscular endurance) and 30-second arm curl test (to assess upper body strength and muscular endurance).
Fatigue | 3-4 months
  Self-reported fatigue will be measured using the Functional Assessment of Cancer Therapy-Fatigue (FACT-F). The FACT-F consists of 13 fatigue-related items and has demonstrated validity and reliability as a brief, standalone measure of fatigue among cancer survivors. The FACT-F will provide a single score, with higher scores indicating better quality of life (QOL) (less fatigue). The FACT-F will be distributed and completed via REDCap at T0 and T1.
Chemotherapy-induced peripheral neuropathy (CIPN) | 3-4 months
  CIPN will be self-reported using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - CIPN-20 item scale. This is a 20-item questionnaire regarding sensory, motor, and autonomic neuropathy symptoms with each item scored from 1 (not at all) to 4 (very much), and all items are summed to result in a score range of 20 to 80. A higher score on the questionnaire indicates more symptom burden from CIPN. Will only administer and score items 1-19 with scores ranging from 16 to 76. This questionnaire will be distributed and completed via REDCap at T0 and T1.
Health-related QOL | 3-4 months
  Will be self-reported using the Functional Assessment of Cancer Therapy-Hepatobiliary questionnaire (FACT-Hep). The FACT-Hep is composed of two parts: the 27-question FACT General (FACT-G) and the 18-question Hepatobiliary Subscale (HS). The FACT-G measures cancer-related QOL in four domains: physical, social/family, emotional, and functional well-being. The HS evaluates the severity of hepatobiliary cancer-specific symptoms. All questions are scored on a Likert scale from 0 to 4 (some are reversed) and added to create FACT-G and HS scores, and these are added to create a FACT-Hep score. A higher FACT-G subscore denotes better QOL. A higher HS subscore denotes a lower degree of disease-related symptoms. The FACT-Hep will be distributed and completed via REDCap at T0 and T1.
Chemotherapy tolerance and delivery | 3-4 months
  Chemotherapy tolerance will be assessed based on relative dose intensities (RDI; defined as the ratio of administered cumulative dose over planned cumulative dose) of the 4 drugs comprising the FOLFIRINOX regimen (39). These data will be collected from participants' electronic health records. Will record if there are any changes in the prescribed regimen (reduction in dose or change in medications) during the study period.
Exercise motivation | 3-4 months
  Will be measured using Behavioral Regulation in Exercise Questionnaire-Version 3 (BREQ-3). The BREQ-3 has subscales measuring external (i.e., performed because of an outside demand or potential reward), introjected (i.e., performed to demonstrate an ability), identified (i.e., consciously valuing exercise), and intrinsic forms of exercise behavior regulation. Participant responses will be evaluated as separate subscale scores and as an overall score, with higher overall scores indicating higher relative autonomy in exercise regulation (i.e., higher personal valuation of exercise and higher intrinsic motivation to exercise). The BREQ-3 will be distributed and completed via REDCap at T0 and T1.
Exercise barriers self-efficacy | 3-4 months
  Participants will complete the Barriers Self-efficacy survey developed by Marcus et al. and adapted by Tirado-Gomez et al. This survey includes 14 questions that assess how confident an individual is in his or her ability to exercise when facing various barriers, such as sickness, fatigue, and lack of time. Participants will indicate their level of confidence using a scale ranging from 1 (not at all confident) to 5 (extremely confident). Responses to the 14 individual items will be summed to obtain an overall score, with a range of 14 to 70.
Social support for exercise | 3-4 months
  Social support for exercise from family and friends will be measured using the Social Support for Exercise Survey (SSES). The SSES lists 13 items that family members or friends may do or say to someone who is trying to exercise regularly, from providing emotional support. The SSES also captures social influences that may hinder exercise. Patients responded to each item separately for friends and family, scoring each item on a Likert-like scale from 1=none to 5=very often. Scores for family and friend participation and family rewards and punishment will be computed following published protocols. Participants will also complete the 13 item scale regarding perceived social support from study interventionists/staff, with instructions to record "does not apply" for items such as "planned for exercise on recreational outings" and "helped plan activities around my exercise." The SSES will be distributed and completed via REDCap at T0 and T1.
Self-reported physical activity | 3-4 months
  Measured using a modified version of the Godin-Shephard Leisure Time Physical Activity Questionnaire (GLTPAQ). The GLTPAQ will be modified as in Vallerand, et al. (2017) to include both aerobic exercise and strengthening exercise related questions and to ascertain performance of guideline-concordant physical activity. To reflect current exercise recommendations, patients will be instructed to include any exercise that lasted at least 5 minutes. Additionally, we will include a single item that asks how many times per week participants perform strengthening exercise (i.e., exercise that improves muscular strength such as weight lifting, resistance bands, sit ups, or push-ups). This question will be extracted from the Health Information National Trends Survey (HINTS) conducted by the National Cancer Institute.
Self-reported physical functioning | 3-4 months
  Self-reported physical functioning will be measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Physical Function 12a. The instrument consists of 12 questions assessing respondents' abilities to perform physical tasks and activities of daily living. Items are scored on 5-point Likert scales, with higher scores indicating higher physical functioning. The PROMIS will be distributed and completed via REDCap at T0 and T1.
Feasibility of Automated Self Assisted 24-hour recall (ASA24) (24-hour dietary recall) | At time of enrollment up to 7-10 days before date of surgery
  Will be assessed by determining the proportion of participants who complete the survey at each target assessment. We will measure the adoption of nutrition recommendations by comparing the recall responses from within the study period to their baseline responses at the time of enrollment. Will also compare adherence to our nutrition recommendations (i.e., protein intake) through the ASA-24 survey at each targeted assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, BA,MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT04837118/ICF_000.pdf